CLINICAL TRIAL: NCT07344103
Title: Association of the Preoperative ROX Index With Early Postoperative Hypoxemia in Adult Patients Undergoing Elective Septorhinoplasty and Endoscopic Sinus Surgery: A Prospective Observational Study
Brief Title: Preoperative ROX Index for Predicting Early Postoperative Hypoxemia in ENT Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, assoc. prof., Istinye University
Other Study IDs: 324-2025
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Hypoxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rox ındex — No intervention; observational study only.

SUMMARY:
Early postoperative hypoxemia is a frequent complication after elective ear, nose, and throat (ENT) surgery and may adversely affect recovery in the post-anesthesia care unit (PACU). Simple and non-invasive preoperative tools to identify patients at risk for early postoperative hypoxemia are limited.

The ROX index, calculated using oxygen saturation, fraction of inspired oxygen, and respiratory rate, is an easily applicable bedside parameter that has been shown to predict respiratory deterioration in various clinical settings. However, its predictive value in the preoperative period for patients undergoing elective ENT surgery has not been well established.

This prospective observational study aims to evaluate the association between the preoperative ROX index measured on room air and early postoperative hypoxemia in adult patients undergoing elective septorhinoplasty or endoscopic sinus surgery under general anesthesia. Early postoperative hypoxemia will be defined as oxygen saturation below 92% or the need for supplemental oxygen at a flow rate of 4 L/min or higher within the first 30 minutes after PACU admission. The predictive performance of the ROX index will be assessed using receiver operating characteristic (ROC) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled for elective septorhinoplasty or endoscopic sinus surgery
* Undergoing surgery under general anesthesia
* Ability to undergo preoperative measurement of oxygen saturation and respiratory rate on room air
* Provision of written informed consent

Exclusion Criteria:

* Age <18 years or >65 years
* ASA physical status III or higher
* Known severe cardiopulmonary disease (e.g., advanced chronic obstructive pulmonary disease, pulmonary hypertension, severe heart failure)
* Active respiratory tract infection in the preoperative period
* Body mass index (BMI) >35 kg/m²
* Requirement for long-term supplemental oxygen therapy
* Refusal or inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 65 years with American Society of Anesthesiologists (ASA) physical status I-II who are scheduled for elective septorhinoplasty or endoscopic sinus surgery under general anesthesia will be included in this study. All participants will undergo standard preoperative assessment, including measurement of oxygen saturation and respiratory rate on room air, and will be monitored postoperatively in the post-anesthesia care unit (PACU) according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Hypoxemia | Within the first 30 minutes after admission to the post-anesthesia care unit (PACU)
  Early postoperative hypoxemia will be defined as an oxygen saturation (SpO₂) below 92% or the requirement for supplemental oxygen at a flow rate of 4 L/min or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Background] Khurshied S, Zahid MA, Babar A, Rafique MH, Khurshid N, Hussain A, Saif M. Effects of Nasal Packing on Patients' Post-operative Vital Signs. Cureus. 2024 Jun 18;16(6):e62616. doi: 10.7759/cureus.62616. eCollection 2024 Jun. PMID 39027799
- [Background] Xiong N, Nong Y, Yi Y. Meta-analysis of risk factors associated with postoperative hypoxemia in the postanesthesia care unit. Am J Transl Res. 2024 Oct 15;16(10):5787-5796. doi: 10.62347/LCKG5157. eCollection 2024. PMID 39544775